CLINICAL TRIAL: NCT05693870
Title: Clinical Evaluation of Different Designs of Fixed Space Maintainer. A Randomized Clinical Trial
Brief Title: Different Designs of Space Maintainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A27080120
Record Dates: First submitted 2023-01-07; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Early Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (B&L) (Experimental): 13 Band and loop (B&L) appliance were included in group one
  Interventions: Device: Fixed space maintainer
- Group II (Ssb&l) (Experimental): 13 Single-sided Band and loop (SsB&L) appliance were included in group two
  Interventions: Device: Fixed space maintainer
- Group III (DBW) (Experimental): 13 Direct Bonded Wire (DBW) appliance were included in group three
  Interventions: Device: Fixed space maintainer
- Group IV(T&L) (Experimental): 13 Tube and Loop (T&L) appliance were included in group four
  Interventions: Device: Fixed space maintainer

INTERVENTIONS:
Device: Fixed space maintainer — Appliance bonded with composite resin or/banded and cemented with glass ionomer cement
  Other Names: Bonded or/ Banded space maintainers

SUMMARY:
Purpose: Evaluation of survival rate for three space maintainers (SMs) of different designs versus standard one.

Methods: 52 extraction sites in children of age group of 4-7 years with prematurely-lost 1st primary molar were selected for this study. The whole sample was divided into four groups (13 each). In Group I, Band and loop (B&L), Group II: Single-sided band and loop (Ss B&L), Group III: Direct bonded wire (DBW), Group IV: Tube and loop (T&L). children were recalled at 3, 6, 9, 12,15-month.

DETAILED DESCRIPTION:
Purpose: Evaluation of survival rate for three space maintainers (SMs) of different designs versus standard one.

Methods: 52 extraction sites in children of age group of 4-7 years with prematurely-lost 1st primary molar were selected for this study. The whole sample was divided into four groups (13 each). In Group I, Band and loop (B&L), Group II: Single-sided band and loop (Ss B&L), Group III: Direct bonded wire (DBW), Group IV: Tube and loop (T&L). children were recalled at 3, 6, 9, 12,15-month. Cumulative survival rates of SMs were estimated by means of Kaplan-Meier method with log rank test. Cumulative survival rates of SMs were estimated by means of Kaplan-Meier method with log rank test. Sample size: The total sample size was calculated using Sampsize application with anticipated success on treatment with conventional band and loop 86% , anticipated response on treatment with direct bonded wire 33% 12, at 80% power, and significant level 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Children and their parents showed cooperation and compliance.
2. Extraction of the first primary molar was not exceeding three months.
3. Angle's class 1 occlusion with normal deciduous molar relation
4. Child not complaining from any systemic disease.
5. The extraction space was of only one missing first deciduous molar with remaining teeth present on mesial and distal side of extraction space.
6. Absence of para-functional habits or abnormal occlusion conditions such as crossbite, open bite, deep bite.
7. No restorative application on the buccal surfaces of abutment teeth, otherwise extra-coronal complete coverage, as stainless-steel crown, was applied only in banded groups.
8. Radiographically, presence of permanent successor.
9. Absence of any pathological evidence on the eruption track of the permanent tooth.
10. Ability to attend follow-up appointments as required.

Exclusion Criteria:

1. Child complaining from any systemic disease.
2. Prescence of para-functional habits or abnormal occlusion conditions such as crossbite, open bite, deep bite
3. Extraction of the first primary molar was exceeding three months.
4. The extraction space resulted from more than one missing deciduous molar
5. Radiographically, absence of permanent successor.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Median survival rate | 15 months
  Cumulative survival rates of space maintainers were estimated by means of Kaplan-Meier method with log rank test

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahem H Elkalla, Professor, Study Director — Department of Pediatric Dentistry Department, Mansoura University, Mansoura, Egypt
Locations (1):
- Department of Pediatric Dentistry, Mansoura University, Al Mansurah, Dakahleya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tunc ES, Bayrak S, Tuloglu N, Egilmez T, Isci D. Evaluation of survival of 3 different fixed space maintainers. Pediatr Dent. 2012 Jul-Aug;34(4):e97-102. PMID 23014081
- [Background] Gulec S, Dogan MC, Seydaoglu G. Clinical evaluation of a new bonded space maintainer. J Clin Orthod. 2014 Dec;48(12):784-90. No abstract available. PMID 25708113
- [Result] Setia V, Kumar Pandit I, Srivastava N, Gugnani N, Gupta M. Banded vs Bonded Space Maintainers: Finding Better Way Out. Int J Clin Pediatr Dent. 2014 May;7(2):97-104. doi: 10.5005/jp-journals-10005-1245. Epub 2014 Aug 29. PMID 25356008
- [Result] Srivastava N, Grover J, Panthri P. Space Maintenance with an Innovative "Tube and Loop" Space Maintainer (Nikhil Appliance). Int J Clin Pediatr Dent. 2016 Jan-Mar;9(1):86-9. doi: 10.5005/jp-journals-10005-1340. Epub 2016 Apr 22. PMID 27274163